CLINICAL TRIAL: NCT00740155
Title: Safety and Immunogenicity of Bivalent and Tetravalent Formulations of Dengue Vaccine Candidates in Healthy Flavivirus-Naïve Adults Aged 18 to 45 Years
Brief Title: Safety and Immunogenicity of Formulations of Dengue Vaccines in Healthy Flavivirus-Naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD11
Record Dates: First submitted 2008-05-07; First posted 2008-08-22 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Dengue Virus; Dengue Fever; Dengue Hemorrhagic Fever; Dengue Diseases
Keywords: Dengue virus; Dengue fever; Dengue hemorrhagic fever; Dengue diseases
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental)
  Interventions: Biological: Bivalent CYD-1,3 Dengue (Vero) + Bivalent CYD-2,4 Dengue (Vero)
- Group 2 (Experimental)
  Interventions: Biological: Bivalent CYD-1,3 Dengue (Vero) + Bivalent CYD-2,4 Dengue (Vero)
- Group 3 (Experimental)
  Interventions: Biological: Tetravalent blending VDV-2/CYD-1,3,4 Dengue (Vero)
- Group 4 (Experimental)
  Interventions: Biological: Tetravalent CYD-1,2,3,4 Dengue (Vero)
- Group 5 (Active Comparator)
  Interventions: Biological: JE-VAX®: Japanese encephalitis virus vaccine inactivated + Tetravalent CYD-1,2,3,4 Dengue (Vero)

INTERVENTIONS:
Biological: Bivalent CYD-1,3 Dengue (Vero) + Bivalent CYD-2,4 Dengue (Vero) — 0.5 mL, Subcutaneous (SC) (CYD-1,3 Day 0; CYD-2,4 Day 105)
  Arms: Group 1
Biological: Bivalent CYD-1,3 Dengue (Vero) + Bivalent CYD-2,4 Dengue (Vero) — 0.5 mL, Subcutaneous (SC) (CYD-1,3 + CYD-2,4 on Day 0 and Day 105)
  Arms: Group 2
Biological: Tetravalent blending VDV-2/CYD-1,3,4 Dengue (Vero) — 0.5 mL, Subcutaneous (SC) (Day 0 and Day 105)
  Arms: Group 3
Biological: Tetravalent CYD-1,2,3,4 Dengue (Vero) — 0.5 mL, Subcutaneous (SC) (Day 0 and Day 105)
  Arms: Group 4
Biological: JE-VAX®: Japanese encephalitis virus vaccine inactivated + Tetravalent CYD-1,2,3,4 Dengue (Vero) — 0.5 mL, Subcutaneous (SC) (JE-VAX® Day 0 + Tetravalent CYD-1,2,3,4 on Day 105)
  Other Names: JE-VAX®
  Arms: Group 5

SUMMARY:
This is part of an ongoing effort to develop a satisfactory dengue vaccine:

Primary objective:

To describe the safety after each vaccination with bivalent and tetravalent formulations of dengue vaccine candidates.

To describe the immune response after each vaccination of dengue vaccine.

DETAILED DESCRIPTION:
Subjects will be randomized to five groups to receive assigned vaccines and followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria :

* Healthy as determined by medical history, clinical examination, and biological safety parameters
* Aged 18 to 45 years on the day of inclusion.
* Informed consent form signed.
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination and at least 4 weeks after the last vaccination.

Exclusion Criteria :

* History of thymic diseases or thymectomy.
* For a woman of child-bearing potential, known or suspected pregnancy or positive pregnancy test
* Breast-feeding
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Human Immunodeficiency Virus (HIV), Hepatitis B (HBs Ag) or Hepatitis C (HC) seropositivity in blood sample taken at screening.
* Laboratory abnormalities considered clinically significant upon the Investigator's judgment or above the intensity thresholds (defined in the protocol) in blood sample taken at screening.
* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Previous residence in or travel of more than 2 weeks to areas with high dengue infection endemicity.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances (i.e. egg, egg products, proteins of rodent or neural origin, gelatin, and thimerosal.
* History of urticaria after hymenoptera envenomation.
* History of flavivirus infection as reported by the subject.
* Previous vaccination against flavivirus diseases (including Japanese encephalitis, tick-borne encephalitis, and yellow fever).
* Planned travel during the present trial period to areas with high dengue infection endemicity.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroid therapy (at a dose of a t least 10 mg).
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past 3 months.
* Any vaccination in the 4 weeks preceding the first trial vaccination.
* Vaccination planned in the 4 weeks following any trial vaccination.
* Flavivirus vaccination planned during the present trial period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety: To provide information concerning the safety of ChimeriVax™ Dengue Vaccine | 12 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Mexico (2):
  - Tlalpan
  - Valle de Chalco

REFERENCES:
- [Result] Dayan GH, Galan-Herrera JF, Forrat R, Zambrano B, Bouckenooghe A, Harenberg A, Guy B, Lang J. Assessment of bivalent and tetravalent dengue vaccine formulations in flavivirus-naive adults in Mexico. Hum Vaccin Immunother. 2014;10(10):2853-63. doi: 10.4161/21645515.2014.972131. PMID 25483647
- See also: Related Info — http://www.sanofipasteur.com